CLINICAL TRIAL: NCT02932319
Title: Outpatient Foley Catheter for Induction of Labor in Nulliparous for Prolonged Pregnancy
Acronym: FOLOUT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Deficient Inclusions
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015_10; 2015-A01298-41 (Other: ID-RCB number, ANSM); PHRCI_2014 (Other: PHRC number, DGOS)
Record Dates: First submitted 2016-10-04; First posted 2016-10-13 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-03

CONDITIONS: Induction of Labour; Prolonged Pregnancy
Keywords: induction of labour; nulliparous; prolonged pregnancy; foley catheter; vaginal birth
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foley catheter (Active Comparator): The patient will have an induction at home after 60 mn of fetal heart rate monitoring.
  Interventions: Device: Foley catheter
- Expectative (Sham Comparator): The patient in this arm will have the actual care (expectative until the next day befor starting the induction)
  Interventions: Other: expectative

INTERVENTIONS:
Device: Foley catheter — The Foley cathter will be inserted at term + 4 days for 24 hours.
  Arms: Foley catheter
Other: expectative — expectative until the next day befor starting the induction
  Arms: Expectative

SUMMARY:
15 to 20 % of nulliparous needs an induction at term. None study has evaluated Foley catheter induction at home versus expectative in this population

ELIGIBILITY:
Inclusion Criteria:

* prolonged pregnancy (D+4) nulliparous no complication during pregnancy location near th hospital (20 mn by car) Bishop < 6

Exclusion Criteria:

* medical history small for gestationnal age PROM Live alone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Bishop score | at term birth +5 days
  Measure the evolution of Bishop score,change between the randomization and the return of the patient

SECONDARY OUTCOMES:
Labour ward | at term birth +5 days
Total dose of prostaglandin used in case of cervical ripening. | During labor
Utilization rate of oxytocin | During labor
Total dose of Ocytocin used or not for induction labor | During labor
number of birth | between the term consultation + 4 days (randomization) and delivery time
delivery rate | within 24 hours and 48 hours after randomization
Caesarean rate | before labor and during labor
Maternal complications | through study completion, at 4 day
  It's the time between the term consultation + 4 days (randomization) and delivery time (day 4)
Fetal complications | through study completion, at 4 day
Neonatal complications | through study completion, at 4 day
Duration of hospital stay | through study completion, at 4 day

CONTACTS AND LOCATIONS:
Overall Officials: Charles Garabedian, MD, Principal Investigator — University Hospital, Lille
Locations (5):
- France (5):
  - CHU de Caen, Caen
  - Hôpital Jeanne de Flandre - CHRU, Lille
  - CH Roubaix, Roubaix
  - CHU Rouen, Rouen
  - Ch Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garabedian C, Tillouche N, Drumez E, Labreuche J, Dreyfus M, Deruelle P. Outpatient balloon catheter versus expectant management for post-term labor induction in nulliparous women: A randomized trial. J Gynecol Obstet Hum Reprod. 2024 Nov;53(9):102822. doi: 10.1016/j.jogoh.2024.102822. Epub 2024 Jul 10. PMID 38997091